CLINICAL TRIAL: NCT01865357
Title: Prospective Longitudinal 1-year Study of the Correlation Between Cognitive Functioning in Patients With Clinically Isolated Syndrome Suggestive of Multiple Sclerosis and Disconnection in the Brain Assessed by MRI:"SCI-COG" Study
Brief Title: Prospective Longitudinal 1-year Study of the Correlation Between Cognitive Functioning in Patients With Clinically Isolated Syndrome Suggestive of Multiple Sclerosis and Disconnection in the Brain Assessed by MRI
Acronym: SCI-COG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: TEVA laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2011/33
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Clinically Isolated Demyelinating Syndromes; Multiple Sclerosis; Cognitive Deficiencies; Brain MRI
MeSH Terms: conditions — Multiple Sclerosis | interventions — Eye Movements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient (Experimental): Clinically isolated neurological syndrome (CIS) compatible with a demyelinating inflammatory episode within the central nervous system, potentially beginning multiple sclerosis (MS) whatever the mode of presentation
  Interventions: Other: Brain MRI - Clinical and cognitive evaluation; Other: Eye movement
- Control (Experimental): healthy subject
  Interventions: Other: Brain MRI - Clinical and cognitive evaluation; Other: Eye movement

INTERVENTIONS:
Other: Brain MRI - Clinical and cognitive evaluation — * Clinical evaluation (EDSS, MSFC)
  * Cognitive evaluation with tests of information processing speed, attention, working memory, episodic memory and executive functions, assessment of confounding factors (depression (BDI) and anxiety (HAD), mood (EHD), fatigue (M-FIS) and assessment of quality of life (SEP-59)
  * Brain MRI (3 Tesla): FLAIR, 3D MPRAGE T1 and DTI
Other: Eye movement — Assessment of eye Movements (EyeBrain software) for only the group of 15 healthy subjects at baseline and at 12 months

SUMMARY:
Clinically isolated demyelinating syndromes (CIS) can evolve into multiple sclerosis (MS). Cognitive deficiencies could occur at this early stage and concern mainly information processing speed (IPS) and their mechanisms are not fully understood. Diffusion Tensor Imaging (DTI) can help in the understanding of these mechanisms.

DETAILED DESCRIPTION:
This is a prospective cohort, observational, longitudinal, monocentric study. This study will include 60 patients with CIS followed for 1 year and 60 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Men and Women
  * ≥16 years
  * Fluent French speaker
  * Clinically isolated neurological syndrome (CIS) compatible with a demyelinating inflammatory episode within the central nervous system, potentially beginning multiple sclerosis (MS) whatever the mode of presentation
  * Between 60 and 180 days from the onset
  * At least two clinically silent lesions on their T2-weighted brain or spinal MRI scan with a size of at least 3 mm, at least one of which being cerebral, ovoid, or periventricular
  * Having a medical insurance
  * Free and informed consent signed
* Controls:

  * Men and Women
  * ≥18 years
  * Fluent French speaker
  * Having a medical insurance
  * Free and informed consent signed

Exclusion Criteria:

* Patients:

  * Prior documented neurological episode suggestive of MS.
  * Other ongoing neurological diseases.
  * Known chronic systemic diseases as judged by the investigator (for instance: lupus, Gougerot-Sjögren, sarcoidosis, sclerodermia, Crohn disease,…).
  * Other causes (trauma, tumor, radiotherapy, infections, vascular diseases, neuromyelitis optica).
  * Current dependence on alcohol or drugs.
  * Dosage change, stop or start of hypnotic or anxiolytic or antidepressive treatment less than 15 days
  * MRI contra-indications.
  * Steroid treatment less than one month (be taken orally or by infusion) at the dosage of 500mg daily.
* Controls:

  * Known chronic psychiatric or neurologic diseases which could interfere with neuropsychological testing, not taking into account stable and mild depressive syndrome
  * Known chronic systemic diseases as judged by the investigator (for instance: lupus, Gougerot-Sjögren, sarcoidosis, scleroderma, Crohn disease…).
  * MS familial history
  * Current dependence on alcohol or drugs
  * Known cognitive impairment
  * Prior neuropsychological testing with the same tests less than one year
  * Dosage change, stop or start of hypnotic or anxiolytic or antidepressive treatment less than 2 months
  * Steroid treatment less than one month (be taken orally or by infusion) at the dosage of 500mg daily.
  * MRI contra-indications
  * Steroid treatment less than one month (be taken orally or by infusion) at the dosage of 500mg daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-08-24 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation between fractional anisotropy (FA) value and cognitive z scores or cognitive impairment indexes for each domains | visit 2 - 1 year after inclusion
  IPS, attention, working memory, episodic memory and executive functions), established by voxel-wise statistics (TBSS) in CIS patients

SECONDARY OUTCOMES:
Comparison of skeleton of FA between CIS patients and healthy subjects | V2 - 1 year after the inclusion
Comparison of cognitive scores at each test between CIS patients and controls | D0 and V2 - 1 year after the inclusion
Proportion of patients with cognitive impairment (≥ 3 tests impaired) and correlations with anxiety, depressive syndrome and fatigue | D0 and V2 - 1 year after the inclusion
Comparison of statistical maps of FA | D0 and V2 - 1 year after the inclusion
  mean cortical thickness and deep grey nuclei volumes with cognitive indexes in the 3 pre-define groups: cognitively preserved CIS patients at baseline and after one year; cognitively impaired CIS patients only after one year and cognitively impaired CIS patients at the two evaluations.
Correlations between cognitive scores and mean cortical thickness and deep grey nuclei volumes in CIS patients | D0 and V2 - 1 year after the inclusion
Comparison of cognitive scores at each test and eye movements scores | D0 and V2 - 1 year after the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BROCHET, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Moroso A, Ruet A, Lamargue-Hamel D, Munsch F, Deloire M, Coupe P, Ouallet JC, Planche V, Moscufo N, Meier DS, Tourdias T, Guttmann CR, Dousset V, Brochet B. Posterior lobules of the cerebellum and information processing speed at various stages of multiple sclerosis. J Neurol Neurosurg Psychiatry. 2017 Feb;88(2):146-151. doi: 10.1136/jnnp-2016-313867. Epub 2016 Oct 27. PMID 27789541